CLINICAL TRIAL: NCT00480168
Title: A Prospective Study to Assess Metabolic Changes in Children and Adolescents Aged 6-18 Treated With Atypical Antipsychotics
Brief Title: A Prospective Study to Assess Metabolic Changes in Children and Adolescents Treated With Atypical Antipsychotics
Status: Completed | Type: Observational
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Sponsor
Other Study IDs: R-05-116; 11172 (Other: REB)
Record Dates: First submitted 2007-05-25; First posted 2007-05-30 (Estimated); Last update posted 2017-08-28 (Actual); Status verified 2017-08

CONDITIONS: Adverse Effects
Keywords: child; adolescent; weight gain; endocrine disruptors
MeSH Terms: conditions — Weight Gain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to observe patients aged 6-18 with various psychiatric diagnosis being treated with drugs called atypical antipsychotics to determine the effects of the drugs on growth, weight gain, and laboratory tests.

DETAILED DESCRIPTION:
Introduction: Antipsychotics have been used for many years to treat serious mental illnesses like schizophrenia and bipolar illness (manic depression). These older drugs carry a higher risk of side effects like shaking, stiffness, restlessness or uncontrolled movements. They may occur when the drugs are first taken, or later, after years of use. Newer drugs called atypical antipsychotics (ATA's) are much less likely to cause these problems. Their lack of these side effects and greater safety have led doctors to use them for other diseases in both adults and younger patients. They have proved to be helpful in aggression, impulsiveness, anxiety and mood swings. Unfortunately, a number of other side effects, such as weight gain, increased rates of diabetes and increases in cholesterol have also been identified. While a lot of current research into these side effects has been done in adults, there have been few studies with younger patients. The research so far has been brief and involved small numbers. This is especially important in this young and potentially vulnerable group of patients.

Study Methods: This research will study children and teens aged 6 to 18 who are being treated with the newer drugs for the first time. If agreeable to the patients and their parents or guardians, their doctors will prescribe one of the newer drugs and will measure the effects, if any, on weight, blood sugar, cholesterol as well as the improvement in their condition. Weight, height, and blood work will be done before the drug is started, and 6 and 12 months after they have been on it, comparing the results with their original values. The doctor, the patient and the parent or guardian will rate the patients' condition at these times, as well, to evaluate their improvement.

ELIGIBILITY:
Inclusion Criteria:

* Atypical Antipsychotic naive patients who have agreed to take Atypical Antipsychotic medication upon the recommendation of their physician based on the child and their symptoms as per their usual patient care
* Outpatients and inpatients
* A wide range of patients including those with ADHD, Tourette's disorder, anxiety, disruptive behavior and mood instability as well as psychosis
* Children and adolescents aged 6 through 18 years
* Both sexes
* Females who have reached menarche and are sexually active who agree to use adequate birth control
* Patients who are willing to give informed assent/consent
* Guardians willing to give informed consent, if needed
* No initiation of or changes of doses of other psychotropic medication prescribed for the indication of which the atypical antipsychotic is being prescribed in the preceding month.

Exclusion Criteria:

* Patients with eating disorders (this condition might affect the expected weight and metabolic changes anticipated with the medications)
* Concurrent medical conditions including diabetes or hyperlipidemia if, in the judgment of the treating physician, the use of atypical anti-psychotics would be contra-indicated. (patient safety)
* Substance abuse (may effect the reliability of the patients or confound weight or metabolic effects of the medications)
* Pregnant or lactating patients (patient safety)

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Community sample of youth 6-18 where treatment with atypical antipsychotic medication is being initiated
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2005-07-05 (Actual); Primary Completion 2012-08-31 (Actual); Study Completion 2012-08-31 (Actual)

PRIMARY OUTCOMES:
Increase in BMI | 12 months

SECONDARY OUTCOMES:
Change in glucose and lipids | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Tamison M Doey, MD FRCPC, Principal Investigator — The University of Western Ontario
Locations (2):
- Canada (2):
  - London Health Science Centre, London, Ontario
  - Windsor Regional Hospital, Windsor, Ontario